CLINICAL TRIAL: NCT04332731
Title: Prairie Renal Denervation Study: Renal Denervation (RDN) for Management of Patients With Loin Pain Hematuria Syndrome (LPHS)
Brief Title: Prairie Loin Pain Hematuria Syndrome Renal Denervation Study: A Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB-17-88
Record Dates: First submitted 2020-03-23; First posted 2020-04-03 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Loin Pain-Hematuria Syndrome
Keywords: Loin Pain; Renal Denervation; Endovascular ablation of renal nerves

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to one of two arms: 1) renal denervation (treatment group) or 2) sham (control group). The experimental group patients will receive a single treatment with radiofrequency ablation applied bilaterally. Similar to the treatment arm, sham patients will be given general anesthesia. The steps will be similar in the sham arm.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The clinical staff (Nephrologist and Nurse) will be blinded to which patients are allocated to the randomized treatment and control groups. Only the interventional radiologist will know at the time of the procedure which group the patient has been assigned to. The radiologist will not be involved with patient follow up following the procedure. This way, the clinical follow-up will not be affected by clinician or patient knowledge of specific patient treatment. Unblinding will occur after the six-month follow-up assessment. The patient will be told the type of treatment received and, if they were allocated to the sham arm, will be offered the opportunity to undergo the RDN procedure. The patient treatment allocation will not be revealed until after the patient's six month follow-up period is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Renal angiography and Renal denervation (Experimental): Symplicity Spyral™ multi electrode renal denervation system
  After renal angiography, participants in the experimental group will be immediately treated with renal denervation procedure using standard techniques. The participants will remain blinded throughout the procedure.
  Interventions: Device: Symplicity Spyral™ multi electrode renal denervation system; Diagnostic Test: Renal angiogram
- Renal angiography (Sham Comparator): In the control group, the sham procedure will consist of only a renal angiogram. Participants will undergo diagnostic renal angiogram but will not receive any therapeutic endovascular treatment. Participants will remain on the procedure table for at least 20 min after the angiogram to prevent possible unblinding of randomization allocation.
  Interventions: Diagnostic Test: Renal angiogram

INTERVENTIONS:
Device: Symplicity Spyral™ multi electrode renal denervation system — Symplicity Spyral™ multi-electrode renal denervation catheter (Symplicity Spyral catheter, Medtronic) and associated Symplicity G3™ renal denervation radiofrequency generator (Symplicity G3 generator, Medtronic) will be used in this study. The Symplicity Spyral™ multi-electrode renal denervation catheter is intended to deliver low-level radio frequency (RF) energy through the wall of the renal artery to denervate the human kidney.
  Other Names: Renal denervation system
  Arms: Renal angiography and Renal denervation
Diagnostic Test: Renal angiogram — Renal angiogram will be used in both treatment and sham groups. Renal angiography is an imaging test used to study the blood vessels in the kidneys. The test will examine the kidney artery anatomy using x-rays following the injection of an x-ray dye (contrast medium). Only patients with eligible renal artery anatomy (between 3 mm and 8 mm) will be randomized ( to treatment or sham groups).
  Other Names: Kidney angiogram

SUMMARY:
Loin Pain Hematuria Syndrome (LPHS) is a poorly understood, painful and incapacitating condition that typically afflicts young women and was first described in 1967. Currently, the treatment for LPHS is opioid prescription and in some extreme cases, surgical denervation of the nociceptive impulses with renal auto transplantation and auto nephrectomy.

Radiofrequency nerve ablation is a minimally invasive alternative to opiate therapy, auto-transplantation and nephrectomy in LPHS. In the investigators' previous exploratory pre/post single centre studies, the investigators showed promising results with regards to pain relief, mood, disability and quality of life post procedure. As these initial studies were neither blinded nor randomized, improvements in pain and quality of life scores owing to a placebo effect cannot be ruled out ; hence, to rule out any cause-effect relation between treatment and outcome, selection-bias, influences the investigators intend to conduct a double-blinded, parallel group, sham-controlled, randomized controlled trial (RCT). The present study is designed to assess the feasibility of conducting a large scale randomized control trial.

Study Hypothesis: In the present study the investigators hypothesize that the recruitment, intervention, measurement and trial procedures will be feasible and acceptable, thus allowing to proceed with a full randomized control trial

DETAILED DESCRIPTION:
Research Design and Methods

This study is a double-blinded, parallel group, sham-controlled, randomized control, partial crossover feasibility trial. This feasibility trial is a part of a larger clinical to trial to assess both statistical and clinical significance of renal denervation treatment in LPHS. This trial will involve 10 Saskatchewan -based patients for whom travel will be covered to and from Regina. These patients will be randomized to either receive the treatment procedure or the sham procedure.

To assess the feasibility measure, the QuinteT recruitment intervention methodology will be utilized, involving a researcher interviewing patients at 6 months after the study (with the inclusion of a satisfaction likert question regarding the study) and interviewing the study personnel throughout the trial. Patient identifiers will be kept anonymous throughout the QuinteT process, and the interviewer will be blind to the treatment allocation of the patient. The feasibility assessments will be reported in accordance with the CONSORT 2010 statement: extension to randomized pilot and feasibility trials guidelines.

The team has produced two manuscripts regarding the impact of renal denervation on LPHS patients. The investigators' initial article outlines four successful case studies reported from a single centre, where "half of the four patients experienced complete pain relief post procedure, whereas the other two patients had a 75% improvement in their frequency of analgesic use" . The investigators then conducted a 12-patient cohort study and observed 10/12 patients at 3 months and 11/12 patients at 6 months reporting a >30% reduction in pain based on the McGill pain questionnaire, along with consistent improvements in disability, mood and quality of life.These results provide the investigators with sufficient preliminary results to scale the hypothesis, improve the study design, and introduce more rigor to the methods so the investigators may use an RCT design to more-definitively assess the effectiveness of renal denervation on pain reduction for LPHS patients.

Trial Intervention:

Renal angiography will be performed to confirm the suitability of renal artery anatomy for renal denervation therapy. If suitability criteria are met, the participant will then be randomized for a sham procedure or a renal denervation procedure. Participants will be randomly allocated to one of two treatment arms: 1) renal denervation (treatment group) or 2) sham treatment (control group) immediately following the renal angiogram. All eligible participants will have an equal chance to be assigned to either treatment or control group with a 1:1 treatment allocation design being used. Participants will be given general anesthesia, thus they will be blinded to their randomized group assignment; they will not know the difference between the renal angiography procedure alone and the renal angiography plus denervation procedure. After the procedure the participants will be sent to the recovery room and the nursing team caring for the patient will be blinded to the procedure. The radiological aspect (sham or procedure) will not be entered on the hospital electronic medical rounds/ PACS. If the angiographic information is needed by other health care professional for a clinical event then it will be released upon request by the Interventional Radiologist.

Treatment Group: Participants remain blinded and are immediately treated with the renal denervation procedure.

Sham Group: Participants remain blinded and remain in the procedure table for at least 20 minutes prior to introducer sheath removal.

Sham Procedure:

In the control group, the sham procedure will consist of only a renal angiogram. Participants will undergo diagnostic renal angiogram but will not receive any therapeutic endovascular treatment. The diagnostic catheter will be kept in situ and dummy radiograph scan will be performed for another 10-15 min before removing the femoral sheath from the sedated patient. Participants will remain on the procedure table for at least 20 min after the angiogram to prevent possible unblinding of randomisation allocation.

The clinical staff (Nephrologist and Nurse Practitioner) and the study coordinator will be blinded to the treatment allocation. Only the interventional radiologist and his/her designated study staff will not be blinded to a participant's randomization group. The radiologist will not be involved with participants follow up following the procedure. This way, the clinical follow-up will not be affected by clinician or participant knowledge of specific treatment. Unblinding will occur after the six-month follow-up assessment. The participant's will be told the type of treatment received and, if they were allocated to the sham arm, they will undergo the RDN procedure. The participant's treatment allocation will not be revealed until after the six month follow-up period is complete. After the initial 6-month follow-up period is over, the participants who were in sham group will undergo the experimental treatment.

Computer software will be used by an analyst, who is not involved with clinical care, to randomly assign patients to either the treatment or control groups. All patients will have an equal chance to be assigned either treatment group with a 1:1 treatment allocation design being used. Currently, the investigators have one site that will treat patients.

Measures

Following measures will be taken at baseline, 6 weeks and 3 and 6 month after the procedure:

EuroQol-5 Dimensions-5 Levels (EQ-5D-5L): A descriptive questionnaire with 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The dimensions have five levels (no, slight, moderate, severe and extreme problems). Participants select the level that corresponds to their perceived health status. Also, there is a vertical visual analogue scale (VAS) from 0 to 100, where participants record their health status lies with the end points being "The worst health the participant can imagine" and "The best health the participant can imagine". The VAS results may be used to quantify the patient's judgement on their own health.

McGill Pain Questionnaire (MPQ): A questionnaire to measure the quality and quantity of patient pain. The scale ranges from no pain (0) to maximum pain (78).

Brief Pain Inventory Questionnaire (BPS): A questionnaire to measure the severity and impact of pain on the patient's daily life and the perceived relief received from current intervention. The short form is has nine-points relating to patients occurrence of pain, areas of pain, rating pain at its worst in the last 24 hours, rating pain at its least in the last 24 hours, average pain level, current pain level, treatments being used, percentage of pain relief form medications used in the past 24 hours and specification of how pain has interfered with life.

Center for Epidemiologic Studies Depression Scale (CES-D): A questionnaire for measuring self-reported depression. Patients are asked to rate over the last week how often they experienced symptoms of depression. Scores range from 0 to 60, with higher score indicating more depression symptoms and lower scores indicating fewer symptoms.

Short Form Health Survey (SF-36): A health-related quality of life questionnaire that elicits information about participants using eight health concepts: physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and mental health. Scores range from 0 to 100, with lower scores relating to more disability and higher scores relating to less disability.

Oswestry Disability Index (ODI): A health questionnaire used to measure patient's functional disability. The questionnaire comprises of ten sections: pain intensity, personal care, lifting, walking, sitting, standing sleeping, sex life, social life and travelling. Index scores range from 0% to 100%, with higher scores relating to more disability and lower scores relating to less disability.

Pain Medication Diary: Participants will be asked to record the number and doses of medications they are taking to alleviate their pain. The type of medication will also be recorded.

SCID-5: A structured assessment tool for DSM-5 disorders (exclusion criteria for the present study). The diagnostic modules can assess somatic symptom disorders, mood disorders, psychotic disorders, substance use disorders, obsessive compulsive and related disorders, anxiety disorders, eating disorders, some sleeping disorders, externalizing disorders and trauma and stress related disorders.

For six weeks and three and six-month assessment the investigators will follow up with the patient, by phone or by in-person visit.

Participant's Follow-up Regimen:

Participants will have the initial treatment of either renal denervation (RDN) or the sham procedure and be followed for 6 months. After this time has elapsed and the treatment allocation is unblinded, participants who received the sham procedure will be given the RDN procedure. Participants will initially have their baseline measurements taken (pain score (MPQ, BPS), quality of life scores (EQ-5D, SF-36), mood (CES-D), and disability (ODI) and then have follow-ups taken at 6 weeks, 3 and 6 months post treatment. Participant's demographic data (Age, gender and race), complete blood count, serum electrolytes, and serum urea/creatinine and urine analysis, BMI and eGFR will also be collected.

Participant's Safety/Discontinuation :

An independent safety committee will be formed to formatively assess risks to patient safety throughout the study. The committee will consist of physicians, researchers and administrators whom are not involved in the study, and have extensive nephrology and/or research experience. The committee will meet before recruitment, upon randomization, bi-weekly during the procedure period, and post-procedure.

Participants are allowed to withdraw from the study at any time without need to explain. Should the independent safety committee report patient safety concerns, the decision will be made as to whether the trial should be discontinued or whether the consent form must be modified to incorporate any new findings, will be made. Should new findings about the efficacy of this procedure for this indication emerge that would impact the premise for the study, the appropriateness of continuing the study will be reviewed. Should an emergency situation occur, the name, ID and treatment allocation of the participant involved in the emergency condition will be given to the principal investigator. The principal investigator will decide if there is an emergency with his experience as a physician. The research team has received biomedical research ethics approval from the former Regina Qu'Appelle Health Region (RQHR), Research Ethics Board.

Statistics:

Analysis for the feasibility trial will be restricted to qualitative thematic analysis and non-parametric analysis to compare the two small patient populations. No power or sample size calculations will be reported as this is not necessary for the feasibility phase of this trial.

ELIGIBILITY:
Inclusion/ Exclusion Criteria

Inclusion criteria for patients to be invited to participate in the study are:

* ≥ 18 years of age
* Diagnosed with loin pain hematuria syndrome by a nephrologist, in consultation with a urologist.
* Current use of prescription pain medication for LPHS treatment
* Arteries with a diameter between 3 mm and 8 mm.

Exclusion criteria for patients to be screened out of the study are:

* History of kidney auto transplantation
* Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m2
* Pregnant or nursing
* Need chronic oxygen support or mechanical ventilation via tracheostomy continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP)
* Renovascular abnormalities
* Prior renal angioplasty, indwelling renal stents and/or aortic stent grafts
* Evidence of a somatoform disorder as per the SCID-5
* Unavailable to travel to Regina, SK one day prior to the procedure to meet with the Principal Investigator and study coordinator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the proportion of participants undergo procedures (treatment or sham) within 6 months | From the start of the study to 6 months after
  We will consider the trial to be feasible if 80% of the target population (10 patients) undergoes procedure (treatment or sham) within 6 months
Assess the of proportion of randomized participants (treatment or control) who entirely complete the follow-up measures | From the date of procedure (for each patient) to 6 months after the procedure
  We will consider the trial to be feasible if 80% of randomized participants (treatment or control) remain in the trial and entirely complete the follow-up measures.

SECONDARY OUTCOMES:
To assess the change from Baseline morphine-equivalent daily dosage of medication at 6 months after procedure (treatment or control) | From the date of procedure (for each patient) to 6 months after the procedure
  We will record and compare the pain medications dosage (milligrams) using pain medication diary at baseline and 6 months after procedure
To assess the change from Baseline McGill Pain score at 6 months after procedure (treatment or control) | From the date of procedure (for each patient) to 6 months after the procedure
  We will record and compare the pain score measured by McGill Pain Questionnaire (0-78) at baseline and 6 months after procedure
To assess the change from Baseline pain severity score_Brief Pain Inventory at 6 months after procedure (treatment or control) | From the date of procedure (for each patient) to 6 months after the procedure
  We will record and compare the pain severity score measured by short form Brief Pain Inventory Questionnaire (0-10) at baseline and 6 months after procedure
To assess the change from Baseline pain interference score _Brief Pain Inventory at 6 months after procedure (treatment or control) | From the date of procedure (for each patient) to 6 months after the procedure
  We will record and compare the pain interference score measured by short form Brief Pain Inventory Questionnaire (0-10) at baseline and 6 months after procedure
To assess the change from Baseline CES-D score at 6 months after procedure (treatment or control) | From the date of procedure (for each patient) to 6 months after the procedure
  We will record and compare the depression score measured by CES-D Questionnaire (0-60) at baseline and 6 months after procedure
To assess the change from Baseline EQ-5D VAS at 6 months after procedure (treatment or control) | From the date of procedure (for each patient) to 6 months after the procedure
  We will record and compare the quality of life scores measured by EQ-5D VAS form (0-100) at baseline and 6 months after procedure
To assess the change from Baseline SF-36 score at 6 months after procedure (treatment or control) | From the date of procedure (for each patient) to 6 months after the procedure
  We will record and compare the quality of life scores measured by SF-36 Questionnaire (0-100) at baseline and 6 months after procedure
To assess the change from Baseline Oswestry Disability Index at 6 months after procedure (treatment or control) | From the date of procedure (for each patient) to 6 months after the procedure
  We will record and compare the diasability scores measured by ODI Questionnaire (0-100%) at baseline and 6 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bhanu Prasad, MD, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Saskatchewan Health Authority, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad B, Giebel S, Garcia F, Goyal K, St Onge JR. Renal Denervation in Patients With Loin Pain Hematuria Syndrome. Am J Kidney Dis. 2017 Jan;69(1):156-159. doi: 10.1053/j.ajkd.2016.06.016. Epub 2016 Aug 12. PMID 27528372
- [Background] Prasad B, Giebel S, Garcia F, Goyal K, Shrivastava P, Berry W. Successful Use of Renal Denervation in Patients With Loin Pain Hematuria Syndrome-The Regina Loin Pain Hematuria Syndrome Study. Kidney Int Rep. 2018 Feb 2;3(3):638-644. doi: 10.1016/j.ekir.2018.01.006. eCollection 2018 May. PMID 29854971
- [Derived] Prasad B, Jafari M, Kour K, Goyal K, Garcia F. Feasibility Study of a Randomized Controlled Trial Investigating Renal Denervation as a Possible Treatment Option in Patients With Loin Pain Hematuria Syndrome. Can J Kidney Health Dis. 2020 Aug 26;7:2054358120951390. doi: 10.1177/2054358120951390. eCollection 2020. PMID 32922827

DOCUMENTS (1):
  • Study Protocol (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04332731/Prot_000.pdf